CLINICAL TRIAL: NCT01739634
Title: The Efficacy of CASAD in Patients With Diarrhea Related to Medullary Thyroid Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salient Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAL 2012-0584
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Diarrhea; Medullary Thyroid Cancer
Keywords: Diarrhea; Medullary thyroid cancer
MeSH Terms: conditions — Diarrhea; Carcinoma, Medullary | interventions — Calcium Aluminosilicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Drug (Experimental): After a 1 week run-in period CASAD will be administered TID for 1 week. Each dose will be 2 500mg CASAD capsules. Patients will be followed for two weeks post active drug administration.
  Interventions: Drug: CASAD

INTERVENTIONS:
Drug: CASAD — CASAD is provided in 500mg capsules.
  Other Names: Calcium Aluminosilicate Anti-Diarrheal.

SUMMARY:
Diarrhea in patients with MTC (Medullary Thyroid Cancer) can be debilitating and, in some cases life threatening. Findings in such patients include volume depletion, renal insufficiency, and electrolyte disorders. Diarrhea can also lead to increased cost of care, reduced quality of life, and treatment delays. Not all patients benefit from conventional anti-diarrheal therapy. CASAD is proven to reduce diarrhea in humans and animals. Clays have water-binding effects, increase the absorptive capacity of the intestinal mucosa, and absorb the excess cytokines which are possible mechanisms of diarrhea in MTC. In this study, we will investigate if starting 1 g CASAD three times a day will ameliorate the severity of diarrhea in patients with MTC. Diarrhea in patients with MTC can be debilitating and, in some cases life threatening. Findings in such patients include volume depletion, renal insufficiency, and electrolyte disorders. We hypothesize that adding CASAD 3 grams/day will reduce the incidence and ameliorate the severity of diarrhea in patients with MTC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medullary thyroid cancer
* Men and women from all ethnic and racial groups
* Diarrhea ( >=3 loose bowel movements per day)
* Duration of diarrhea of at least 1 week

Exclusion Criteria:

* Patients with MEN 2b (since these patients may have megacolon)
* Patients taking any clay products
* History of significant neurological or psychiatric disorders that would impede giving consent, treatment, or follow up.
* Patients who cannot comply with medications
* Patients whose current medication schedule would not permit an approximate 2 hour window between administration of CASAD and other scheduled medications.
* Pregnancy or lactation
* Patients receiving systemic chemotherapy (includes tyrosine kinase inhibitors)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy in treatment of diarrhea | 1 week
  To evaluate the efficacy of CASAD 3 grams per day in reducing the severity of diarrhea after 1 week of treatment in patients with MTC.

SECONDARY OUTCOMES:
Functional impact of CASAD | 1 week
  To explore the functional impact of CASAD and the relative impact of diarrhea in relation to other symptom issues using MDASI-THY (M.D. Anderson Symptom Inventory-Thyroid, appendix D)
Effect on thyroid function tests | 1 week
  To explore the effect of CASAD on thyroid function tests, thyroid hormone and calcium absorption
Changes in MDASI-THY scores | 1 week
  To examine changes in MDASI-THY scores after treatment with CASAD

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States